CLINICAL TRIAL: NCT01053026
Title: Evaluation of Vascular Function, Effects of Exercise Training and Angiotensin Receptor II Antagonist in Patients With Type II Diabetes and Hypertension by Using Near-infrared Spectroscopy, Rapid Laser Doppler Blood Flow Imaging and Circulating Biomarkers
Brief Title: Evaluation of Effects of Exercise Training and ARB in DM Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Daiichi Sankyo Taiwan Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 200903006R
Record Dates: First submitted 2010-01-18; First posted 2010-01-21 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-07

CONDITIONS: Vascular Function; Exercise Training
Keywords: Angiotensin receptor II antagonist
MeSH Terms: interventions — olmesartan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: olmesartan — (1) Olmesartan treatment or (2) Life modification and exercise training

SUMMARY:
The aims of this clinical trial are to assess the impacts on vascular function tests and circulating biomarkers of a short-term (12-week) low-to-median intensity exercise training or ARBs treatment in patients with DM and hypertension.

DETAILED DESCRIPTION:
Inclusion criteria: type II diabetic and hypertensive patients who are aged 30 to 70 year-old with HbA1c ≤ 8.0 % and systolic blood pressure ≥ 140 mmHg. Neither ACEI nor ARB is administrated in recent 6 months. None has significant concomitant systemic diseases such as active infection, malignancy, hepatic or significant renal dysfunction at the time of enrollment (i.e. total bilirubin > 3 mg/dl，ALT > 2.5 times the upper limit of normal range and creatinine > 3 mg/dl in our hospital). Information regarding smoking, hypertension, hyperlipidemia as well as history of cardiovascular disease is obtained from all subjects. No other medication will be modified during the study period. After enrollment, patients are assessed to (1) olmesartan (20 mg per day, with titration), (2) life modification/exercise training for 12 weeks. Vascular function and exercise capacity studies, and peripheral blood testing are performed at baseline and at 12- week follow-up. Data are collected as mean ± SD showing comparison between groups by use of 2-sample t test and chi-square analysis for continuous and categorical variables, respectively. Adjust for the HbA1c level will be adjusted using simple adjustment method (ANCOVA or equivalent regression analysis) while doing the data analysis. Changes between baseline and follow-up measurements are assessed by paired t test. The frequencies of adverse effects between groups will also be comparing by 2-sample t test. A p value <0.05 is defined as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with diabetes mellitus and hypertension
* age 30-70 years，systolic blood pressure 140-160 mmHg and HbA1c ≤ 8%,
* no history of ACEI or ARB use within 6 months

Exclusion Criteria:

* active cardiovascular diseases
* severe hepatic
* renal dysfunction (CRE ≥ 3 mg/dl，T-Bil ≥ 3 mg/dl)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diabetes melitus and hypertension
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
1. Vascular function testing | 12 weeks

SECONDARY OUTCOMES:
Exercise capacity testing | 12 weeks
Circulating biomarkers including hs-CRP, adiponectin, myostatin, MMP, etc | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Wen Wu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan